CLINICAL TRIAL: NCT04828902
Title: Incidence of Postoperative Delirium After Cardiac Surgery in Adults - a Prospective Observational Cohort Study
Brief Title: Incidence of Postoperative Delirium After Cardiac Surgery in Adults.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Maciej M. Kowalik, MD, PhD, Promotor, Dr hab. n. med. Maciej Michał Kowalik, Medical University of Gdansk
Other Study IDs: NKBBN/4421/2020
Record Dates: First submitted 2021-03-21; First posted 2021-04-02 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Delirium; Adult Cardiac Surgery; Covid19
Keywords: postoperative delirium; cardiac surgery; Covid19
MeSH Terms: conditions — Emergence Delirium; COVID-19 | interventions — Cardiac Surgical Procedures; Coronary Artery Bypass; Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac surgery — Any heart surgery on or without cardiopulmonary bypass performed under general anesthesia in the Cardiac Surgical Department, Medical University of Gdańsk.
  Other Names: cabg; valve surgery; aorta surgery; heart transplant; other cardiac surgery

SUMMARY:
Postoperative delirium is an acute syndrome of mental deterioration characterized by acute onset and fluctuating course during the day. Very frequent delirium is a presage of other serious comorbidities i.e.: sepsis, acute kidney injury, circulatory and/or respiratory failure. A detailed knowledge of symptoms and early diagnose of delirium increase the chances of early therapy. To what extent the occurrence of postoperative delirium influences hospital therapy in the Cardiac Surgical Postoperative ICU in University Clinical Centre in Gdańsk is unknown so far.

DETAILED DESCRIPTION:
Study type: prospective, observational cohort study. Facility: tertiary, university hospital Methods: Patients will undergo routine, continuous observation for symptoms of delirium by a trained nursing staff. Occurrence of delirium, Delirium Observation Screening Scale (DOSS) grading, and therapy will by annotated on case record forms (CRFs) every 12 hours. Additionally, collected will be known risk factors of delirium: schedule type, age, arterial hypertension, atrial fibrillation, body mass index (BMI), angiotensin converting enzyme (ACE) inhibitors / angiotensin receptor blockers (ARBs) therapy, hearing loss, dementia, peripheral artery disease, myocardial infarction, depression, diabetes, corona virus disease 2019 (COVID19) infection and/or vaccination; and outcome data: hospital-LOS, prolonged sedation, antipsychotic therapy, surgical reintervention, hours on mechanical ventilation (HOV), number of tracheal intubations, length of consciousness disorders, blood product transfusions, cardiopulmonary resuscitation (CPR), renal replacement therapy (RRT), mechanical circulatory support (MCS), duration of catecholamine support, ICU readmissions, new antibiotic therapies, 30-day mortality.

Statistical methods: Delirium morbidity and risk will be calculated from two-by-two table. Associations between delirium and secondary outcome measures will be evaluated by simple and logistic regression with use of ANOVA test for continuous variables with homogeneous distribution, or Kruskal-Wallis test for continuous variables with non-homogeneous distribution, or categorical variables. Significant will be considered results with p<0.05.

A period of one year was assumed sufficient to draw conclusions on the primary endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 y.a.), undergoing cardiac surgery, who will sign an informed consent to participate in the study.

Exclusion Criteria:

* Deny to sign or absence of an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender will be reported as declared by the subjects.
Study Population: All adult patients undergoing elective/emergency cardiac surgery will be considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Delirium incidence and risk | Through hospitalisation in Postop-ICU - an average of 2 days
  Incidence and risk of postoperative delirium
Risk factors of delirium. | Through hospitalisation in Postop-ICU - an average of 2 days
  collected will be known risk factors of delirium: schedule type, age, arterial hypertension, atrial fibrillation, BMI, ACE/ARBs therapy, hearing loss, dementia, peripheral artery disease, myocardial infarction, depression, diabetes, COVID19 and/or vaccination for it; and outcome data: hospital-LOS, prolonged sedation, antipsychotic therapy, surgical reintervention, direct coercion, length of mechanical ventilation, number of tracheal intubations, length of consciousness disorders, blood product transfusions, cardiopulmonary resuscitation, renal replacement therapy, mechanical circulatory support, duration of catecholamine support, ICU readmissions, new antibiotic therapies, 30-day mortality.
Association between delirium and length of stay in ICU (LOS-ICU). | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and length of stay in ICU (LOS-ICU).

SECONDARY OUTCOMES:
DOSS | Through hospitalisation in Postop-ICU - an average of 2 days
  Associations between delirium and mean DOSS
Hospital-LOS | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and hospital-LOS
Prolonged sedation, antipsychotic therapy and surgical re-intervention. | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and prolonged sedation, antipsychotic therapy, surgical reintervention.
Hours on ventilator. | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and HOV.
Intubations | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and number of tracheal intubations.
Consciousness disorders | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and length of consciousness disorders.
Transfusions | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and blood product transfusions.
CPR, RRT, MCS | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and CPR, RRT, and MCS.
Catecholamines | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and duration of catecholamine support.
ICU readmissions | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and ICU readmissions.
New antibiotic | Through hospitalisation in Postop-ICU - an average of 2 days
  Association between delirium and new antibiotic therapy.
30-day mortality | 30 days after operation
  Association between delirium and 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Lango, Prof.dr.hab., Study Chair — Medical University of Gdańsk, Department of Cardiac Anesthesiology; Maciej Kowalik, Dr hab., Study Director — Medical University of Gdańsk, Department of Cardiac Anesthesiology; Pawel Kozak, Mgr. Piel., Principal Investigator — Medical University of Gdańsk, Department of Cardiac Anesthesiology
Locations (1):
- Department of Cadiac Anesthesiology, Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized patients data are planned to be uploaded into a public data repository (ZENODO.com) after data completion.